CLINICAL TRIAL: NCT03094429
Title: An Adaptive Phase II/III, Double-Blind, Randomized, Placebo-controlled, Two-Part, Dose-Finding, Multi-center Study of the Safety and Efficacy of NaBen®,a D-Amino Acid Oxidase Inhibitor, as an Add-on Therapy With Clozapine, for Residual Symptoms of Refractory Schizophrenia in Adults
Brief Title: An Adaptive Phase II/III, Two-Part, Double-Blind, Randomized, Placebo-controlled, Dose-Finding, Multi-center Study of the Safety and Efficacy of NaBen®, as an Add-on Therapy With Clozapine, for Residual Symptoms of Refractory Schizophrenia in Adults
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SyneuRx International (Taiwan) Corp (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNR-05
Record Dates: First submitted 2015-11-16; First posted 2017-03-29 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Refractory Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NaBen® - 2000 mg/day (Active Comparator): Two NaBen® ( 500 mg) will be taken twice daily at a total dose of 2000 mg/day during this study.
  Interventions: Drug: NaBen®
- NaBen® - 1000 mg/day (Active Comparator): One NaBen® (500 mg) and one placebo will be taken twice daily at a total dose of 1000 mg/day during this study.
  Interventions: Drug: NaBen®
- Placebo - 0 mg/day (Placebo Comparator): The control treatment is placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NaBen® — 2000 mg/day or 1000 mg/day, twice daily
  Arms: NaBen® - 1000 mg/day; NaBen® - 2000 mg/day
Other: Placebo — 0 mg total, twice daily
  Arms: Placebo - 0 mg/day

SUMMARY:
This is an adaptive, Phase II/III study in 2 parts (i.e. Part 1 (dose ranging) and Part 2 (Hypothesis testing)). NaBen® is granted Breakthrough Therapy Designation by US FDA as treatment for refractory schizophrenia.

Part 1 Objectives: There are two primary objectives for Part 1 of this study:

1. To evaluate, in terms of dose-response, the effectiveness of NaBen® (1000 and 2000 mg/day) compared to Placebo (0 mg/day), when combined with clozapine, in improving the residual symptoms associated with refractory schizophrenia in adults, and; to determine the optimal dose to be used in Part 2 of this study.
2. Sample size re-assessment to evaluate the final sample size needed to proceed with Part 2 of the study The secondary objective of the Part 1 of this study is to evaluate the safety and tolerability of NaBen® (1000 and 2000 mg/day) compared to Placebo (0 mg/day), in combination with clozapine.

Part 2 Objectives: The primary objective of the Part 2 of this study is to evaluate the effectiveness of NaBen® (at the optimal dose determined in the Part 1 of this study) compared to Placebo (0 mg/day), when combined with clozapine, in improving the residual symptoms associated with refractory schizophrenia in adults. The secondary objective of the Part 2 of this study is to evaluate the safety and tolerability of NaBen® (at the optimal dose determined in the Part 1 of this study) compared to Placebo (0 mg/day), in combination with clozapine.

DETAILED DESCRIPTION:
This is a Phase II/III, double-blind, randomized, placebo-controlled, two-part, dose-finding, Multi-center study, in which subjects with refractory schizophrenia will be enrolled.

This study will be conducted in two parts:

In Part 1 (i.e. dose finding portion) of the study One hundred seventy one (171) subjects will be randomized in a 1:1:1 ratio (NaBen® 2000 mg/day: NaBen® 1000 mg/day: Placebo).

All subjects, after signing the Informed Consent Form (ICF), will be assessed during the screening phase. This screening phase is designed to exclude subjects who have had more than 20 percent reduction in the PANSS total score using PANSS score evaluations at Visit 1 and Visit 2. Only those subjects who successfully complete the screening phase and still meet the study eligibility criteria will proceed with Randomization and the double-blind treatment. All randomized subjects will receive eight (8) weeks of randomized treatment (NaBen® 2000 mg/day, NaBen® 1000 mg/day or Placebo). Study treatments will be given twice daily.

An Interim Analysis (IA) will be conducted when 171 subjects in Part 1 of the study have been randomized and completed 8 weeks of treatment or early terminated, whichever occurs first. Randomization of subjects in the study will continue until the IA of the Part 1 data is completed. The data from the Part 1 analysis will be reviewed by an independent Data Safety and Monitoring Committee (DSMC) who would assess the data for both safety and efficacy trends. The DSMC responsibilities will be further elaborated in the DSMC charter. The DSMC will approve continuation of the study and recommend the optimal dose and sample size adjustment for the Part 2 of the study.

Assuming no sample size adjustment was made as a result of the IA, for Part 2 of the study a total of 116 subjects will be randomized in a 1:1 ratio, of which 58 subjects will be randomized to the NaBen® optimal dose group and 58 subjects to the Placebo group. The procedures and assessments for subjects in Part 1 and Part 2 of this study will be identical with the exception of the randomization schema.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are between 18 and 55 years of age inclusive
2. Subject is capable of providing informed consent and is willing to sign the ICF prior to study Screening and agrees to comply with the study protocol requirements, or the subject has a Legally Authorized Representative (LAR) who can provide consent to be enrolled into the study
3. If female and not infertile (defined below), the subject must agree for the duration of the study to use one of the following forms of contraception 1) systemic hormonal treatment 2) an Intrauterine device (IUD) which was implanted at least 2 months prior to screening or 3) "double-barrier" contraception (condom, diaphragm and spermicide are each considered a barrier). Females are considered to be infertile if they are either a) surgically sterile or b) have had spontaneous amenorrhea for at least the last 2 years and at least 2 years after the onset of amenorrhea while not receiving hormone replacement therapy and had a Follicle-Stimulating Hormone (FSH) level greater than 40 mIU/mL and an estradiol level less than 30 pg/mL
4. The subject has Physician confirmed DSM-V diagnosis of schizophrenia for the past 2 years based on subject's recorded history and confirmed by psychiatric evaluation and MINI International Neuropsychiatric Interview For Schizophrenia and Psychotic Disorders, version 7.0 (MINI, Version 7.0)
5. The subjects should have refractory schizophrenia as defined below (should meet at least two: either a and b; or a and c; or a and b and c):

   1. Prior non-response to at least 2 antipsychotic drugs of two different chemical classes for at least 4-6 weeks each at doses ≥ 400 mg equivalents of chlorpromazine or 4 mg/day risperidone, AND
   2. No period of good functioning in previous 2 years; OR,
   3. Moderate to severe psychopathology (total PANSS score equal or more than 70): including persistent psychotic symptoms, recurrent mood symptoms, repeated suicide attempts or suicidal ideation, uncontrolled aggressive behavior, moderate to severe positive or negative symptoms or moderate-severe cognitive impairment
6. The subject has been receiving clozapine for a minimum of 6 months with the dose range of 200-900 mg/day. The dose should have remained unchanged for at least 3 months prior to Screening and not expected to change during the study
7. The subject is outpatient, and has been consistently symptomatic without significant fluctuation per the Investigator, with no hospitalization for worsening of schizophrenia within 3 months of the Screening. If the subject is hospitalized during the study for worsening of schizophrenia symptoms the subject will be withdrawn from the study
8. The subject has a minimum PANSS total score of 70 at the Screening and Baseline Visits (Visits 1 and 2)
9. Without clinically significant abnormalities in physical exam, neurological exam and laboratory assessments (urine/blood routine, biochemical tests and ECG) which would exclude the subject from the study in the opinion of the Investigator. For ALT and AST, clinically significant is defined as above two and a half times the upper limit of normal
10. Body Mass Index (BMI) between 17 and 38 inclusive
11. Subject has a negative routine urine illicit drug screening test (including heroin, amphetamines (including MDMA/ecstasy), cocaine, cannabis or PCP)
12. The subject has a caregiver or some other identified responsible person (e.g., family member, social worker, caseworker, or nurse) as determined by the Investigator and per the local regulations. The identified caregiver should be considered reliable by the Investigator and per the local regulations in providing support to the subject to help ensure compliance with study treatment, study visits and protocol procedures who preferably is also able to provide input helpful for completing study rating scales
13. The subject must not be a danger to themselves or others per the Investigator's judgment

Exclusion Criteria:

1. Meets the DSM-V criteria at Screening for intellectual disability, dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, schizophreniform disorder, autistic disorder, primary substance-induced psychotic disorder, dementia, or any other comorbid mental disorders that in the opinion of the Investigator may interfere with study conduct and results interpretation
2. Initiation or dose change of lithium, antidepressant or other mood stabilizers within 16 weeks prior to Screening
3. Initiation or dose change of benzodiazepines or sleep medications, or any other psychotropic medications due to worsening of schizophrenia symptoms or medication side effects within four (4) weeks prior to Screening
4. The subject has previously received NaBen®
5. History of epilepsy, major head trauma, or any neurological illness other than Tourette's syndrome which might impair the subject's cognition or psychiatric functioning per the Investigator's judgment
6. History of allergic reaction to sodium benzoate
7. Serious medical illnesses such as end-stage renal disease, liver failure or heart failure that, in the opinion of the Investigator, may interfere with the conduct of the study
8. Any significant gastrointestinal disorders that, in the opinion of the Investigator, markedly alter the absorption, metabolism or elimination of sodium benzoate
9. Any movement disorders with a total score higher than 6 on SAS scale, or more than 2 on any items of the AIMS scale
10. Current substance abuse, or history of meeting criteria for moderate or severe substance abuse (including alcohol, but excluding nicotine and caffeine) in the past six (6) months prior to Screening
11. Female subjects who are pregnant (as confirmed by serum pregnancy test performed at Screening Visit) or are breast feeding
12. History of cancer not in remission for the last three (3) years except for basal cell carcinoma and squamous cell carcinoma
13. Participation in a clinical trial within 3 months prior to Screening or more than two clinical trials within 12 months
14. Electroconvulsive Therapy (ECT) within 6 months prior to Screening
15. The subject started a new non-medication treatment for schizophrenia or other psychiatric condition within the last 3 months prior to Screening (e.g. individual psychotherapy, cognitive behavioral therapy or rehabilitative therapy)
16. The subject's anti-EPS medications dose or regimen has changed within 2 weeks prior to Screening
17. The subject's PANSS total score has decreased more than 20 percent using PANSS score evaluations at Visit 1 and Visit 2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 287 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | 8 weeks after randomized treatment
  Mean change from baseline in Positive and Negative Syndrome Scale (PANSS) total score

SECONDARY OUTCOMES:
Percent change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | 8 weeks after randomized treatment
  Percent change from baseline in PANSS total score treatment
Percentage of subjects with 20% or more reduction from baseline in Positive and Negative Syndrome Scale (PANSS) total score | 8 weeks after randomized treatment
  Percentage of subjects with 20% or more reduction from baseline in PANSS total score after treatment
Percent change in PANSS sub-scales and Marder PANSS factor scores | 8 weeks
  Percent change in PANSS sub-scales and Marder PANSS factor scores
Percent change in Personal and Social Performance (PSP) scale | 8 weeks
  Percent change in Personal and Social Performance (PSP) scale
Percent change in Schizophrenia Quality of Life Scale (SQLS) | 8 weeks
  Percent change in Schizophrenia Quality of Life Scale (SQLS)
Percent change in Clinical Global Impression-Severity (CGI-S) and -improvement (CGI-I) | 8 weeks
  Percent change in Clinical Global Impression-Severity (CGI-S) and -improvement (CGI-I)
Percent change in Hamilton Depression Rating Scale (HDRS) | 8 weeks
  Percent change in Hamilton Depression Rating Scale (HDRS)
Serum pharmacokinetic evaluations-Maximum Plasma Concentration [Cmax] | 8 weeks
  Serum pharmacokinetic evaluations-Maximum Plasma Concentration [Cmax]
Serum pharmacokinetic evaluations-Area Under the Curve [AUC] | 8 weeks
  Serum pharmacokinetic evaluations-Area Under the Curve [AUC]

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAE) and incidence of withdrawals from the study due to TEAEs | 8 weeks
  Incidence of TEAE and incidence of withdrawals from the study due to TEAEs
Percent change in Simpson-Angus extrapyramidal side effects Scale (SAS) | 8 weeks
  Percent change in Simpson-Angus extrapyramidal side effects Scale (SAS)
Percent change in Abnormal Involuntary Movement Scale (AIMS) | 8 weeks
  Percent change in Abnormal Involuntary Movement Scale (AIMS)
Percent change in Barnes Akathisia Rating Scale (BARS) | 8 weeks
  Percent change in Barnes Akathisia Rating Scale (BARS)
Assessment of suicidality per the Columbia-Suicide Severity Rating Scale (C-SSRS) | 8 weeks
  Assessment of suicidality per the Columbia-Suicide Severity Rating Scale (C-SSRS)
Changes and shifts in laboratory measurements-Hematology | 8 weeks
  Changes and shifts in laboratory measurements-Hematology
Changes and shifts in laboratory measurements-Biochemistry | 8 weeks
  Changes and shifts in laboratory measurements-Biochemistry
Changes and shifts in laboratory measurements-Urine analysis | 8 weeks
  Changes and shifts in laboratory measurements-Urine analysis
Changes in vital signs-Body temperature (°C) | 8 weeks
  Changes in vital signs-Body temperature (°C)
Changes in vital signs-Heart rate (beats per minute) | 8 weeks
  Changes in vital signs-Heart rate (beats per minute)
Changes in vital signs-Respiration rate (breaths per minute) | 8 weeks
  Changes in vital signs-Respiration rate (breaths per minute)
Changes in vital signs-Blood pressure (mm Hg) | 8 weeks
  Changes in vital signs-Blood pressure (mm Hg)
Changes in BMI (in Weight (kg) / [Height (m)]2) | 8 weeks
  Changes in BMI (in Weight (kg) / [Height (m)]2)
Changes in Electrocardiogram (ECG) | 8 weeks
  Changes in Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact SyneuRx International Corp., Pasadena, California, United States